CLINICAL TRIAL: NCT02978950
Title: SToP: Venous Thromboembolism Screening in the Trauma Population
Acronym: SToP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1050048
Record Dates: First submitted 2016-11-23; First posted 2016-12-01 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Venous Thromboembolism; Deep Vein Thrombosis; Trauma, Multiple
Keywords: duplex ultrasound; trauma; venous thromboembolism; prevention
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Multiple Trauma; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surveillance arm (Experimental): Bilateral duplex ultrasound surveillance
  Interventions: Other: Duplex ultrasound surveillance
- No surveillance arm (Active Comparator): no duplex ultrasound surveillance
  Interventions: Other: No ultrasound surveillance

INTERVENTIONS:
Other: Duplex ultrasound surveillance — bilateral lower extremity venous duplex
  Arms: Surveillance arm
Other: No ultrasound surveillance — will have daily exam and history as per normal clinical routine
  Arms: No surveillance arm

SUMMARY:
This is a prospective, randomized vanguard trial of trauma patients admitted to the trauma surgery service at Intermountain Medical Center who are deemed to be at high risk for venous thromboembolism. Once identified and enrolled, subjects will be randomized to receive bilateral lower extremity duplex ultrasound surveillance versus no surveillance. The study will compare the two groups with regard to deep vein thrombosis, pulmonary embolism, and major and clinically relevant bleeding episode rates, both during the index hospitalization and at 90 days post-discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatient status on Intermountain Medical Center (IMC) trauma surgery service, admitted within 24 hours of injury.
2. Age ≥18 at the time of injury
3. Meets the definition of high-risk for VTE according to current IMC trauma service guidelines

Exclusion Criteria:

1. Patient age <18 years at the time of admission to the hospital
2. Pregnancy
3. Prisoners
4. Patients with a life expectancy of less than 30 days
5. Patients with a known hypercoagulable state including:

   * Factor V Leiden
   * Protein C and S deficiencies
   * Dysfibrogenemia of any sort
   * Active cancer
   * Antiphospholipid antibody syndrome
   * History of DVT or PE within past 6 months
   * Myeloproliferative disorders
6. Patients on therapeutic anticoagulation who do not have their agent held upon admission to the hospital.
7. Patient elects to opt-out of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Asymptomatic lower extremity DVT | during index hospitalization, up to 2 weeks
  any DVT found in the lower extremity

SECONDARY OUTCOMES:
Symptomatic DVT propagation from calf veins to proximal veins | 14 days from hospital discharge
  calf vein clot that moves to popliteal vein or higher
Symptomatic/fatal pulmonary embolism | 90 days from hospital discharge
  any pulmonary embolism diagnosed by computed tomography angiogram
Major and clinically relevant bleeding episodes | during index hospitalization, up to 2 weeks
  as defined by the International Society of Thrombosis and Hemostasis
Composite outcome of proximal DVT plus major and clinically relevant bleeding episodes | during index hospitalization, up to 2 weeks
  additive outcome of above knee thrombosis plus major and clinically relevant bleeding
All cause mortality | 90 days
Symptomatic DVT | 90 days
  any lower extremity thrombosis that causes clinical symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Majercik, MD,MBA, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kay AB, Morris DS, Woller SC, Stevens SM, Bledsoe JR, Lloyd JF, Collingridge DS, Majercik S. Trauma patients at risk for venous thromboembolism who undergo routine duplex ultrasound screening experience fewer pulmonary emboli: A prospective randomized trial. J Trauma Acute Care Surg. 2021 May 1;90(5):787-796. doi: 10.1097/TA.0000000000003104. PMID 33560104

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT02978950/Prot_SAP_000.pdf